CLINICAL TRIAL: NCT00070759
Title: Daclizumab for Active, Non-infectious, Sight-threatening Uveitis: A Phase II Pilot Study
Brief Title: Daclizumab to Treat Non-Infectious Sight-Threatening Uveitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040006; 04-EI-0006
Record Dates: First submitted 2003-10-07; First posted 2003-10-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-10-02

CONDITIONS: Uveitis
Keywords: Daclizumab; Uveitis; Active; Acute
MeSH Terms: conditions — Uveitis; Motor Activity | interventions — Daclizumab

INTERVENTIONS:
Drug: Daclizumab

SUMMARY:
This study will examine the safety and effectiveness of treating uveitis, an eye inflammation, with a monoclonal antibody called daclizumab. Monoclonal antibodies are genetically engineered proteins made in large quantities and directed against a specific target in the body. Daclizumab is designed to prevent a specific chemical interaction needed for immune cells called lymphocytes to produce inflammation. In an ongoing NIH study of 10 adults with uveitis, 8 patients were able to decrease corticosteroids and other immunosuppressive medicines they were taking while receiving daclizumab for months or even years. Seven patients continue to take the drug.

Patients 18 years of age and older with active non-infectious intermediate or posterior uveitis in both eyes who require treatment for their disease may be eligible for this study. Candidates will be screened with the following tests and procedures:

* Medical history and physical examination.
* Eye examination to measure visual acuity and eye pressure, and examine the lens, retina, pupils and eye movements.
* Blood tests to measure the number and types of blood cells.
* Fluorescein angiography to check for abnormalities of eye blood vessels. A yellow dye injected into an arm vein travels to the blood vessels in the eyes. Pictures of the retina are taken with a special camera that flashes a blue light into the eye. The pictures show if any dye has leaked from the vessels into the retina, indicating possible abnormalities.

Participants come to the NIH Clinical Center for treatment and follow-up visits. The first daclizumab treatment is given as a 90-minute infusion through a vein. A second IV infusion is given 7 days later. If the treatment has successfully reduced the eye inflammation after 2 weeks, then subsequent treatments are given through injections under the skin once a month for up to 1 year. Patients whose eye disease is not improved after 2 weeks stop the study treatments and receive alternative therapy.

Follow-up visits are scheduled 7, 14, and 21 days after enrollment and at each treatment visit to evaluate the response to treatment and drug side effects. During these visits, patients repeat the exams done at screening. Extra blood samples are taken at certain visits to measure blood levels of daclizumab and to perform clinical laboratory and immunology tests. Fluorescein angiography is done at enrollment and after 1 year.

DETAILED DESCRIPTION:
Uveitis refers to intraocular inflammatory diseases that are an important cause of visual loss. Standard systemic immunosuppressive medications used for uveitis can cause significant toxic side effects, especially with prolonged use. Consequently, an effective treatment with a safer side effect profile is highly desirable. Daclizumab is a humanized monoclonal antibody directed against the high affinity IL-2 receptor CD25 or Tac subunit. The IL-2 receptor system plays a central role in mediating immune responses. Blocking this system impedes immune responses and can inhibit local inflammatory responses, including uveitis. Pilot studies using intravenous or subcutaneous daclizumab treatments suggest that daclizumab treatments at 1 mg/kg every 2-4 weeks for quiescent uveitis may effectively replace the other immunosuppressive medications in a majority of cases.

Because we have little experience using daclizumab for active uveitis, this feasibility study will enroll five study participants that would normally be treated with systemic, high-dose corticosteroids or other cytotoxic, systemic immunosuppressive medications. Since daclizumab for other indications can be tolerated with repeated dosing at 8-10 mg/kg, we will administer daclizumab to reach high serum levels with a pair doses at 8 mg/kg and 4 mg/kg two weeks apart. The primary objective of this study is to collect preliminary information on the utility of acute daclizumab therapy on active ocular inflammation. The primary outcome is resolution of active disease defined as the reduction of vitreous haze by at least 2 steps (from 2+ to Trace, or 1+ to none) and is assessed at 21 days after the initial daclizumab injection. Secondary outcomes will include fluorescein retinal vascular leakage, CME, anterior chamber cells, and visual acuity. In addition all adverse events will be collected regardless of possible relation to daclizumab. Participants who show a 2 step reduction in vitreous haze at day 21 will be permitted to continue SC daclizumab maintenance treatments beginning at Day 28 at 2 mg/kg every 4 weeks for a year. At any time during the followup period, if a participant loses greater than 3 lines of visual acuity from baseline study treatments will be discontinued.

ELIGIBILITY:
* INCLUSION CRITERIA:

Volunteers will be considered eligible participants for this study provided they meet all of the following inclusion criteria:

1. Participant has a diagnosis of active, non-infectious intermediate or posterior uveitis, which may include but is not restricted to the following conditions known to cause intermediate or posterior uveitis: panuveitis, intermediate uveitis of the pars planitis subtype, sarcoidosis, the Vogt-Koyanagi-Harada (VKH) syndrome, birdshot retinochoroidopathy, retinal vasculitis and sympathetic ophthalmia;
2. Participant has active uveitis with greater than or equal to Grade 1 (1+) vitreous haze in at least one eye including evidence of retinal vascular leakage using fluorescein angiography or the presence of cystoid macular edema (CME) at enrollment;
3. Participant's uveitis is currently treated or untreated at the time of enrollment;
4. Participant has best-corrected distance visual acuity (BCVA) in the worst eye of 20/400 or better (ETDRS logMAR less than 1.34);
5. Participant does not plan to undergo elective ocular surgery (e.g., cataract extraction) during the study period;
6. Participant, male or female, with reproductive potential and who is sexually active agrees to use double-barrier contraception methods throughout the course of the study (minimum of 52 weeks) and for 6 additional weeks after completion of the protocol treatment period.

EXCLUSION CRITERIA:

A volunteer will not be permitted to enroll if they meet any one of the following exclusion criteria:

1. Participant is under 18 years of age;
2. Participant has received previous treatment with an IL-2 or IL-2R directed therapy within the past 90 days;
3. Participant has lens opacities or obscured anterior ocular media upon enrollment such that reliable evaluation and grading of posterior segment cannot be performed (except that anterior chamber cells due to inflammation is not an exclusion);
4. Participant has a history of an active herpes zoster or varicella infection within 6 weeks before enrollment, or chicken pox exposure within 21 days before enrollment.
5. Participant has a known history of HIV infection;
6. Participant is currently enrolled in another investigational or interventional therapeutic trial, or is using a therapy for a non-uveitis condition that would likely affect immune responses or interfere with trial logistics, or has received any investigational therapy within the 30 days prior to enrollment;
7. Participant has a history or diagnosis of Behcet's disease (since subsequent tapering or withdrawal of concomitant immunosuppressive medications is not a standard-of-care for Behcet's patients) or a primary diagnosis of anterior uveitis (e.g., HLA-B27 associated uveitis, or ocular conditions usually treated with local and not systemic medications);
8. Participant has a significant local or systemic infection requiring medical treatment at the time of enrollment;
9. Participant is currently pregnant or lactating;
10. Participant has a history of cancer (other than a non-melanoma skin cancer or in situ cervical cancer) diagnosed within the past 5 years;
11. Participant has a non-ocular, medically significant co-morbid condition that impairs normal activities, requires immunosuppression, or has a condition with a prognosis that indicates a significant risk of disability or death if the condition were to continue or be exacerbated during the study period, or a medical condition that would likely have an impact on the participant's ability to comply with the visit schedule. Such conditions may include, for example, recent heart attack, significant COPD, brittle diabetes, kidney disease, severe emphysema, organ transplant (requiring corticosteroids or other immunosuppressive medications), hepatitis or other liver disease, or uncontrolled psychiatric illnesses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6
Dates: Start 2003-10-06; Study Completion 2006-10-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Lacomba MS, Martin CM, Chamond RR, Galera JM, Omar M, Estevez EC. Aqueous and serum interferon gamma, interleukin (IL) 2, IL-4, and IL-10 in patients with uveitis. Arch Ophthalmol. 2000 Jun;118(6):768-72. doi: 10.1001/archopht.118.6.768. PMID 10865312